CLINICAL TRIAL: NCT07068737
Title: The Effect of a Structured Bathing Care Package on Comfort and Skin Hydration in Preterm Infants in the Neonatal Intensive Care Unit
Brief Title: Effect of a Bathing Care Package on Comfort and Skin Moisture in Preterm Infants in a Neonatal Intensive Care Unit
Acronym: NICU-BATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kiymet Aygün (Other)
Responsible Party: Sponsor-Investigator, Kiymet Aygün, Principal Investigator BSc, MSc Kıymet Aygün, Tarsus University
Organization: Tarsus University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NICU-BATH-2025
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Preterm Birth; Skin Hydration in Preterm Infants; Comfort in Neonates; Bathing Care Package; Neonatal Nursing Care
Keywords: newborn; bath; bundle; nursing
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: There is a bath care package group and a group that undergoes routine bathing at the clinic (control group). Randomisation was not performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bathing care package group (Experimental): bathing care package group
  Interventions: Behavioral: bathing care package
- routine bath group (Active Comparator): routine bath group
  Interventions: Behavioral: routine bath

INTERVENTIONS:
Behavioral: bathing care package — Participants receive a bathing care package that includes a swaddled immersion bath. Room temperature is maintained at 26-27°C with 40-60% humidity. Bath water temperature is controlled at 37-38°C. The infant is swaddled and immersed in water up to the shoulders while the head remains above water. The bath lasts no longer than 5 minutes. After bathing, the infant is gently dried without rubbing, wrapped in a towel, and placed in a pre-warmed incubator (31-34°C) for 10 minutes.
  Arms: Bathing care package group
Behavioral: routine bath — Participants receive routine bathing care according to NICU standards. This includes hand hygiene before the procedure, preparing necessary materials, placing the infant in a mesh sling in the bath, washing the body from clean to dirty areas with soft sponges and hospital-provided cleansing agents. The bath lasts up to 10 minutes. After bathing, the infant is quickly dried without rubbing and then diapered.
  Arms: routine bath group

SUMMARY:
This completed study evaluated the effects of a bathing care package on the comfort level and skin hydration of preterm infants admitted to the neonatal intensive care unit (NICU). Preterm infants, born before 37 weeks of gestation, often experience skin dryness and discomfort due to their immature skin barrier.

The bathing care package involved a gentle bathing procedure using warm water at a specific temperature, performed in a basin with a wrapping technique. This procedure was carried out under controlled room temperature and humidity conditions to maximize infant comfort. Comfort-enhancing techniques were also applied during and after the bath.

Preterm infants were randomly assigned to either the intervention group receiving the bathing care package or the control group receiving the standard bathing care routinely practiced in the NICU.

Data collected throughout the study demonstrated that the bathing care package helped maintain skin hydration and preserve comfort levels better than the standard care.

The findings contribute to improving neonatal nursing protocols aimed at enhancing the well-being of preterm infants.

All procedures were conducted with informed consent from parents or legal guardians and approved by the institutional ethics committee.

DETAILED DESCRIPTION:
Background: The first bath of a baby admitted to the Neonatal Intensive Care Unit (NICU) is usually performed in the neonatal intensive care environment. Preparing the intensive care environment before bathing is very important for the newborn's adaptation. Preterm infants, in particular, are more sensitive to stressors encountered during nursing care that negatively affect their neurodevelopment. Bathing is an application that increases comfort in preterm infants, but it is also an application that causes a stress response, so it is important to make bathing less stressful and more comfortable. Bathing is performed using different methods. Studies have shown that the swaddling bath method, one of these methods, increases comfort and reduces stress in preterm infants compared to other methods and better maintains body temperature.

The epidermal barrier begins to form during intrauterine life and continues to develop after birth. The skin of a preterm infant is immature compared to that of a term infant and is still developing. The hydration and moisture of the stratum corneum layer are indicators of skin barrier function and prevent transepidermal water loss (TEWL). In preterm infants, due to inadequate stratum corneum formation, there is a risk of transepidermal water loss and impaired skin barrier function . High transepidermal water loss values indicate that the skin barrier is weakened and allows more water to evaporate from the body. This can lead to dehydration and increased sensitivity to external irritants and pathogens. Low transepidermal water loss values indicate that the skin barrier is functioning well, effectively retaining moisture and protecting against environmental factors . Bathing is a practice that increases skin moisture and protects the skin barrier.

Aim: This study was conducted because there was no existing study in our country that simultaneously examined the effects of skin moisture and comfort levels in preterm infants due to the absence of a standardised care package application that combines optimal bathing conditions. In this study, a bathing care package was developed to increase the comfort level and skin moisture of preterm infants.

Methods: The study was conducted as a pre-test and post-test controlled semi-experimental design. Data were collected using the "Information Form", "Newborn Comfort Scale", and "Follow-up Form". A skin moisture measuring device, bedside monitor, liquid temperature gauge, and room temperature and humidity measuring devices were used to collect data. The study was initiated after obtaining ethical approval and clinical permission. Parents of preterm infants in the control group and the group receiving the care package who met the inclusion criteria were informed about the study, and their written consent was obtained. The study was conducted in the neonatal intensive care unit of a city and teaching research hospital. The sample size was calculated using the "G. Power-3.1.9.2" programme. The effect size was calculated as 0.926, with a 95% confidence interval and 95% power, requiring a total of 64 preterm newborns, with at least 32 in each group.

First, the data for the control group were collected. The control group underwent bathing according to the clinic's routine practice.

The clinic's routine bathing practice: Hands are washed according to hand hygiene rules before the procedure. Before bathing, the tub and water in which the baby will be bathed, a mesh bag appropriate for the baby's size, a towel for drying, cleaning materials for body cleansing, and a baby diaper are prepared. To prevent the baby's body temperature from dropping, doors and windows that create air currents in the room are closed. A mesh is stretched over the tub and the baby is laid on it. The baby is washed from clean to dirty, keeping the midline position, by wetting the arms and shoulders and pouring the washing material provided by the hospital onto a soft disposable surgical cap, lathering it, and rinsing it with water from a bucket. The same procedure is applied to the abdomen, genital area, feet, and legs. Finally, the baby's head is washed, and the bath is completed. The bathing process is completed within 10 minutes. After the bath, the baby is quickly wrapped in a towel. The baby's body is gently dried without rubbing. The baby's nappy is changed.

The care package to be used in the study was prepared. The appropriateness of the care package, prepared in accordance with the literature, was reviewed by seven experts in the field (nurses, doctors, faculty members).

Nurses were trained on the bathing procedure using slides based on the contents of the bathing care package. The training was conducted by the same person.The bath care package contains the necessary materials for bathing and the steps for bathing. In addition, the researcher filmed a video showing these steps. The video was shown to nurses after each training session. The researcher observed that the steps for bathing were being followed correctly. The effectiveness of the application was observed by the researcher. In addition, posters were hung in patient rooms so that nurses could check the accuracy of the application steps during bathing.

Data was collected from the group to which the care package was applied. Bathing was initiated in accordance with the care package.

Contents of the bathing care package applied:

The room temperature is maintained at 26-27°C, and the humidity at around 40-60%. The bath water temperature is measured using a thermometer that measures liquid temperature and is maintained at 37-38°C. The immersion bath method, in which the baby is swaddled (in a cradle), is used to better maintain body temperature and vital signs . After the baby is swaddled, the head and shoulders are placed on the arm and supported while maintaining the flexed and midline position. The lower extremities are immersed first, followed by the abdominal region, and finally the shoulders. The water in the tub should cover the baby's body up to the shoulders, with the head remaining above the water . Each time, a different part of the baby's body is washed, starting from the cleanest to the dirtiest. The eyes are wiped from the inside out with a damp, soft gauze pad, and a separate pad is used to clean the face. The arms and shoulders are washed, followed by the abdomen, genital area, feet, and legs. Finally, the head is washed to complete the bath. The bath should not last longer than five minutes . After the bath, the baby is quickly wrapped in a dry towel. The baby is placed in a dry incubator at a temperature of 31-34°C and kept wrapped for 10 minutes. The baby's body is not rubbed dry. After 10 minutes, the baby is diapered.

The vital signs of preterm babies before and after bathing were measured, including body temperature, heart rate, respiratory rate, oxygen saturation (SPO2), skin moisture, and comfort. The nurse assessed the vital signs (body temperature, heart rate, respiratory rate, oxygen saturation (SPO2)), skin moisture, and comfort score of the infant at 15 and 30 minutes before and after the bath and recorded them in the monitoring form.

ELIGIBILITY:
Inclusion Criteria:

* Parental consent to participate in the study
* Gestational age between 32 and 37 weeks
* Admission to the Neonatal Intensive Care Unit
* Spontaneous breathing
* Stable physiological parameters
* Birth weight above 1500 g
* 24 hours have passed since birth (WHO)

Exclusion Criteria:

* Birth weight below 1500 g
* Dependence on mechanical ventilation
* Diagnosed with sepsis
* Receiving sedatives and/or muscle relaxants
* Chromosomal abnormality
* Infant of a mother with hepatitis or HIV
* Meconium aspiration
* Chest tube, central venous catheter, drain, peritoneal dialysis catheter.

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-05-04 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Neonatal comfort score | Before bath, and at 15 and 30 minutes after bath
  The comfort level of preterm infants will be assessed using the Neonatal Comfort Behavior Scale (NCBS) at baseline and at 15 and 30 minutes after bathing to determine whether the bathing care package helps maintain comfort.
  Each item on the scale is scored from 1 to 5, and the evaluation is based on the total score. The total score on the Neonatal Comfort Behavior Scale (NCBS) can range from a minimum of 6 to a maximum of 30. A total score between 14 and 30 indicates that the infant is experiencing pain or distress, is not comfortable, and requires interventions to promote comfort.
Skin moisture level | Before bath, and at 15 and 30 minutes after bath
  Skin moisture levels of preterm infants will be measured using a non-invasive skin hydration monitor before the bath, and at 15 and 30 minutes after bathing to evaluate the effect of the bathing care package on skin moisture retention.

CONTACTS AND LOCATIONS:
Overall Officials: Kıymet Aygün, MSc, Principal Investigator — Tarsus University
Locations (1):
- Mersin City Education and Research Hospital, Mersin, Toroslar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the vulnerable nature of the study population (preterm infants) and ethical considerations regarding privacy and confidentiality. Institutional policies also restrict public data sharing.